CLINICAL TRIAL: NCT04132193
Title: Correlation of Musicality and Cognitive Skills in Persons With Alzheimer´s Disease
Brief Title: Processing of Music in Alzheimer Patients
Acronym: MUKU-DEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Seppo Soinila, professor, chief physician, Turku University Hospital
Other Study IDs: T112/2019
Record Dates: First submitted 2019-10-08; First posted 2019-10-18 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease; Dementia; Amusia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Correlation of musicality, brain atrophy in brain areas relevant for music processing and the stage of Alzheimer´s disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia accounting for 60-70% of all dementias. In most cases the cause for AD is unknown. The progression of AD is characterized by an advancing decline in cognitive skills and symptoms like impaired learning, memory deficits, language impairment and behavioral disturbances in later stages. The symptoms of AD are caused by cerebral atrophy which is the consequence of multiple pathological processes, including the formation of neurofibrillary tangles at neurites and amyloid plaques in the walls of cerebral blood vessels. AD is a major public health issue and its significance increases as the population grows older.

Music is thought to have preceded the development of spoken language as a form of communication and it has been used for therapeutic purposes in many ways throughout history. In patients with AD, musical memory has been noticed to be well-preserved and constituting a relatively independent part of memory. Music-based neurological rehabilitation provides a mode of treatment, which is free of side effects and can be personalized for patients with dementia.

Aims of this study are to examine how AD affects the structure of various brain areas associated with music processing and to statistically correlate musical cognition with memory performance in patients with AD. Focus is on brain areas associated with musical pleasure like the striatum, superior temporal gyrus, inferior frontal gyrus and areas associated with long-term musical memory like the anterior cingulate gyrus and presupplementary motor area. Hippocampal atrophy serves as a reference of the stage of AD. Our working hypothesis is that musicality correlates with preserved cognitive skills and memory.

Voluntary participants who have been diagnosed with AD are recruited from Turku University Central Hospital. Their musicality is assessed with a short version of Montreal Battery of Evaluation of Amusia which contains listening tasks that test the patients' memory, rhythm recognition and pitch discrimination. In addition, patients are asked to fill an inquiry that maps their use of music and its significance in their daily lives. Voxel-Based Morphometry is applied on MRI images to evaluate atrophy in the hippocampus and entorhinal cortex, which correlate with clinical stages of AD, as well as on the brain areas relevant for processing of music.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed Alzheimer´s disease

Exclusion Criteria:

Other neurological comorbidity, substance abuse

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of Southwest Finland Hospital District
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Montreal Battery of Evaluation of Amusia | 60 minutes
  Number of correct answers in three task collections (total 79 tasks)
Brain atrophy in MRI scans | 120 minutes
  Loss of volume in brain regions relevant for music processing and in the hippocampi estimated by voxel-based morphometry
CERAD (Consortium for Establishing Registry of Alzheimer´s Disease) | 30 minutes
  Level of cognitive impairment

SECONDARY OUTCOMES:
Use of music in patient´s daily life | 30 minutes
  Validated self-report questionnaire MusEQ in Finnish, Likert scale 1-5 (Vanstone AD et al, Aging Ment Health 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Soinila, MD PhD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No